CLINICAL TRIAL: NCT00318695
Title: Influence of Probiotics on Prevention of Atopy, Atopic Disease and Immunological Responses- A Randomized Double-Blind Placebo Controlled Trial
Brief Title: Influence of Probiotics on Prevention of Atopy, Atopic Disease and Immunological Responses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SQNU01
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Eczema; Asthma; Allergic Rhinitis
Keywords: Probiotics; Eczema; Asthma; Allergic Rhinitis; Prevention; Immunological responses
MeSH Terms: conditions — Eczema; Asthma; Rhinitis, Allergic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): Bifidobacterium longum [BL999] and Lactobacillus rhamnosus [LPR]
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Commercially available cow's milk based infant formula without probiotic supplementation
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Bifidobacterium longum [BL999] and Lactobacillus rhamnosus [LPR]
  Arms: Probiotics
Other: Placebo — Commercially available cow's milk based infant formula without probiotic supplementation
  Arms: Placebo

SUMMARY:
This will be a double-blind, randomized placebo-controlled study. 253 children were recruited and randomly assigned into one of 2 groups to receive either normal infant formula or formula with Bifidobacterium longum and Lactobacillus rhamnosus GG. The primary aim is to assess the effect of early administration (from birth) of probiotics on the incidence of allergic sensitization, eczema, asthma and rhinitis.

DETAILED DESCRIPTION:
One of the most important early influences on the immune system is the intestinal microflora. The gastrointestinal tract, being the largest body area interacting with the environment, is one of the earliest to be colonized and is quantitatively the most important source of microbial stimulation for the immature immune system. Probiotics are helpful bacteria from healthy intestinal tract, and have shown potential in reducing allergy. This is extremely important as allergic diseases are on the rise worldwide. Probiotics are safe, easy to administer and can be used early for intervention as allergic sensitization, once established, is difficult to reverse.

This double-blind, randomized placebo-controlled study has recruited 253 children from birth. These babies, with a family history of atopic disease, will be randomly assigned into one of 2 groups to receive either normal infant formula or formula with Bifidobacterium longum and Lactobacillus rhamnosus GG. The formula will be consumed postnatally for 6 months, after which the child will continue with normal follow-on milk. Children will be examined at the neonatal period and at 1, 3, 6, 12 and 24 months. Blood samples will be collected at birth (cord blood) and at 1 year of age. Blood will be analyzed for cytokines, total IgE and specific IgE. Skin prick test for common allergens will also be performed at 1 year of age. Stools will be collected at 5 days, 1, 3, 12 months and analyzed for the pattern of stool colonization.

ELIGIBILITY:
Inclusion Criteria:

* Parents agree to the subject's participation in the study and informed consent has been obtained.
* Either parent or sibling (i.e. first degree relative) has a history of atopy. This will be evidenced by a doctor-diagnosis of asthma, allergic rhinitis or eczema and a positive skin prick test to any of a panel of common allergens.
* The subject is born at above 35 weeks of gestation and weighs above 2 kg.
* The subject does not have major congenital malformations/major illness.
* Family appears to be able to successfully complete this trial.

Exclusion Criteria:

* Mother has a medical illness, which in the opinion of the investigator, will interfere with the results of the study.
* The parent is unable/unwilling to comply with procedures.
* The parents choose to totally breast-feed the child.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2004-05; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Atopic eczema by 2 years of age

SECONDARY OUTCOMES:
Asthma by 2 years of age
Allergic Rhinitis by 2 years of age
Allergen sensitization by 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lynette Shek, Consultant, Principal Investigator — National University Hospital (NUH), Singapore
Locations (1):
- National University Hospital (NUH), Singapore, Singapore